CLINICAL TRIAL: NCT01279486
Title: Clearblue Home Pregnancy Test Consumer Study
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-0187
Record Dates: First submitted 2010-12-24; First posted 2011-01-19 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-01

CONDITIONS: Pregnancy
Keywords: Pregnancy,

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Approximately 120 female volunteers requesting a pregnancy test will be recruited locally to the UK trial centre.

Volunteers will be required to use the Clearblue Pregnancy Test according to the product instructions, and provide a urine sample from the same void.

Trained technicians will conduct a second test from the urine sample.

DETAILED DESCRIPTION:
Approximately 120 female volunteers attending the study site requesting a pregnancy test will be recruited locally to the UK trial centre.

Volunteers will be required to use the Clearblue Pregnancy Test according to the product instructions, and provide a urine sample from the same void.

Trained technicians will conduct a second test from the urine sample to evaluate performance between consumer and technician testing.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 year old
* Female
* Requesting a pregnancy test

Exclusion Criteria:

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers requesting a pregnancy test
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanagaratnam Shanmugaratnam, Principal Investigator — National Health Service, United Kingdom
Locations (2):
- United Kingdom (2):
  - Bedford General Hospital, Bedford, Bedfordshire
  - Brook clinic, Milton Keynes

IPD SHARING:
Plan to Share IPD: No
Overview will be available after study is completed

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnancy Test: Volunteers were instructed to carry out the pregnancy test according to the instruction leaflet and collect a urine sample from the same void into the provided urine container. Volunteers were told to conduct the test according to the instruction leaflet. No other instructions were given. Volunteers were free to choose the "in-stream" or "dip" method of sampling.
Period: Overall Study
Arm/Group | Pregnancy Test
Started | 120
Completed | 119 (1 result questionnaire was not returned so 119 volunteers results were used for consumer accuracy.)
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All volunteers were actively seeking a pregnancy test.
Arm/Group | Pregnancy Test
Number analyzed (Participants) | 120
Age, Customized [Count of Participants; unit: Participants]
  Age: 18-25 | 96
  Age: 26-30 | 11
  Age: 31-35 | 5
  Age: 36-40 | 5
  Age: 41-45 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 8
  Race/Ethnicity: Black or African American | 15
  Race/Ethnicity: Native Hawaiian or other Pacific Islander | 0
  Race/Ethnicity: White | 94
  Race/Ethnicity: American Indian or Alaska Native | 0
  Race/Ethnicity: Mixed | 3
Educational Status [Count of Participants; unit: Participants]
  Degree, or equivalent, and above | 12
  Other higher education below degree level | 13
  A levels, vocational level 3 and equivalents | 31
  GCSE (grade A*-C), vocational level 2 and equivale | 45
  Qualifications at level 1 or below | 2
  Other qualifications | 5
  No qualifications | 10
  Unclear | 2
Occupation [Count of Participants; unit: Participants]
  Managerial | 7
  Professional | 10
  Associate Professional / Technical | 0
  Administrative / Secretarial | 7
  Skilled Trade | 0
  Personal Services | 1
  Sales / Customer Services | 21
  Manufacturing / Driver | 1
  Support Personnel | 0
  Student | 29
  Homemaker | 14
  Other | 28
  Unclear (ticked more than one category) | 2

OUTCOME MEASURES:

1. Primary Outcome: Consumer Agreement
Description: The agreement of the consumer Clearblue Pregnancy Test result with technician Clearblue Pregnancy Test results when testing the same sample.
Time Frame: During testing approximately 15 minutes
Population: 2 volunteers were not included due to insufficient sample. Another volunteer had a error result and there was insufficient sample to repeat.
Measure: Number; unit: percentage of agreement
Arm/Group | Pregnancy Test
Number analyzed (Participants) | 117
percentage of agreement | 100

ADVERSE EVENTS:
Time Frame: Duration of study (December 2010 - June 2011). Each volunteer presented to the study site for 1 hour maximum.
Arm/Group | Pregnancy Test
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes